#### **RESEARCH CONSENT FORM**

# In-Depth Interview with Health Service Staff: CONSENT FORM EVALUATION OF OPENSRP IN ZAMBIA

# **Evaluating the Efficacy of Using a Digital Consumption Management Tool for Family Planning in Zambia**

PI: Veronika J Wirtz, BPharm, PhD

Email: vwirtz@bu.edu

NCT 05503992

Date: 10/07/2022

**RESEARCH CONSENT FORM** 

In-Depth Interview with Health Service Staff: CONSENT FORM

**EVALUATION OF OPENSRP IN ZAMBIA** 

**Background** 

**Purpose** 

We would like to speak with you because you are either a CHW or a staff member at a district or health facility involved in this study. We want to understand your perceptions on family planning services in this area, barriers and facilitators to implementing family planning programs in rural communities here, and recommendations on how to improve these programs/systems. For those involved in using the OpenSRP mobile application, we would also like to know barriers and facilitators to use and recommendations for improving the application.

What Happens in this Research?

You will be one of approximately 112 participants asked to complete this qualitative interview. The overarching study will take place in 40 health facility catchment areas in Zambia from four districts in Luapula Province.

If you agree to take part, we will ask you questions about perspectives on family planning commodities stock, tracking, and distribution systems, relevant training received, barriers and facilitators to implementation of these systems, and perceptions of the OpenSPR system compared to standard processes (if applicable). This interview will take no longer than 1 hour.

During the interview, notes will be taken on what is said. If you agree, we will also audio-record the discussion to make sure that we do not miss what is said. We will write down your first name for this study, but we will keep it private. When we write reports from this discussion, we may show what you say, but we will never use your name at any time.

Risk and Discomforts

The risk of taking part in this study is that other people may hear what you say. It is important that you not share anything that you are not comfortable sharing. You do not have to respond to any question unless you feel comfortable doing so. We can stop at any time if you need to.

**Potential Benefits** 

You will receive no direct benefits from your participation in this study. However, your participation may help us better understand how to improve stocking and distribution of family planning commodities in this district.

**Alternatives** 

You can choose not to take part in the study. If you decide not to take part or withdraw from the study, you will not suffer any penalties or lose any benefits or services to which you are entitled.

**Participant Costs and Payments** 

There are no costs to you for participating. You will not be paid to participate in this study.

IRB NUMBER: H-43082

2

## **RESEARCH CONSENT FORM**

#### In-Depth Interview with Health Service Staff: CONSENT FORM

**EVALUATION OF OPENSRP IN ZAMBIA** 

## **Confidentiality**

We will keep your name and answers private. Your interview will be assigned a number. Your information will be kept in the locked file, only study team members can see these data. When the information is published, we will not link what you said to your name.

# **Participants Rights**

By consenting to participate in this study, you do not waive any of your legal rights. Giving consent means you have heard or read the information about this study and that you agree to participate. You will be given a copy of this form to keep.

You may obtain further information about your rights as a research participant by contacting the ERES Converge Research Ethics Committee at +260977493220. The investigator or a member of the research team will try to answer all your questions. If you have questions or concerns at any time, please contact Dr. Lloyd Matowe +260972547447 or, if he is not available, you can contact the Program Manager Mr. Paul Kango at +260973172281. You can also contact the ERES Converge Research Ethics Committee at +260977493220 or Boston University Medical Campus Institutional Review Board at +16173585372.

# Rights to Refuse or Withdraw

Taking part in this study is voluntary. You have the right to refuse to take part. If you decide to take part in the study and then you change your mind, you can withdraw from the research. Your participation is completely up to you. If you choose to take part, you can stop at any time. If there are any new findings during the study that may affect whether you want to continue to take part, you will be told about them as soon as possible.

The investigator may decide to discontinue your participation without your permission because he/she may decide that staying in the study will be bad for you, or the sponsor may stop the study.

By signing below, you are agreeing to participate which indicates that you have read this consent form or have had it read to you, that your questions have been answered to your satisfaction, and that you voluntarily agree to participate in this research study. You may keep the copy of this for your records.

| Name of participant: | Date: |
|---------------------------------------|-------|
| Thumbprint/ Signature of participant: | |
| Name of witness: | Date: |
| Signature of witness: | |